CLINICAL TRIAL: NCT02276378
Title: Influence of Food on the Bioavailability of Telmisartan 40 mg/HCTZ 12.5 mg Fixed-dose Combination and of Telmisartan 80 mg/HCTZ 12.5 mg Fixed-dose Combination in Japanese Healthy Male Volunteers (an Open-label, Randomised, Single-dose, Two-way Crossover Study)
Brief Title: Influence of Food on the Bioavailability of Two Doses of Telmisartan/HCTZ Fixed-dose Combination in Japanese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.569
Record Dates: First submitted 2014-10-27; First posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Hydrochlorothiazide

ARMS (4):
- Telmisartan low / HCTZ fixed-dose combination, fed (Experimental)
  Interventions: Drug: Telmisartan low; Drug: Hydrochlorothiazide (HCTZ); Other: Japanese meal
- Telmisartan high / HCTZ fixed-dose combination, fed (Experimental)
  Interventions: Drug: Telmisartan high; Drug: Hydrochlorothiazide (HCTZ); Other: Japanese meal
- Telmisartan low /HCTZ fixed-dose combination, fasted (Active Comparator)
  Interventions: Drug: Telmisartan low; Drug: Hydrochlorothiazide (HCTZ)
- Telmisartan high /HCTZ fixed-dose combination, fasted (Active Comparator)
  Interventions: Drug: Telmisartan high; Drug: Hydrochlorothiazide (HCTZ)

INTERVENTIONS:
Drug: Telmisartan low
  Arms: Telmisartan low / HCTZ fixed-dose combination, fed; Telmisartan low /HCTZ fixed-dose combination, fasted
Drug: Telmisartan high
  Arms: Telmisartan high / HCTZ fixed-dose combination, fed; Telmisartan high /HCTZ fixed-dose combination, fasted
Drug: Hydrochlorothiazide (HCTZ)
Other: Japanese meal
  Arms: Telmisartan high / HCTZ fixed-dose combination, fed; Telmisartan low / HCTZ fixed-dose combination, fed

SUMMARY:
To investigate the relative bioavailability and pharmacokinetics of the fixed-dose combination tablets (telmisartan 40 mg/HCTZ 12.5 mg and telmisartan 80 mg/HCTZ 12.5 mg) after food intake in comparison with those in the fasting state in healthy Japanese male volunteers

ELIGIBILITY:
Inclusion Criteria:

Healthy males according to the following criteria:

1. Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR), body temperature), 12-lead ECG (electrocardiogram), clinical laboratory tests
2. Age ≥20 and Age ≤35 years
3. Body weight ≥50 kg
4. BMI ≥18.0 and BMI ≤25.0 kg/m2 (Body Mass Index)
5. Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation.

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
3. Chronic or relevant acute infections
4. Any clinical relevant findings of the laboratory test deviating from normal
5. Positive result for either hepatitis B surface (HBs) antigen, anti Hepatitis C virus (HCV) antibodies, syphilitic test or human immunodeficiency virus (HIV) test
6. History of surgery of gastrointestinal tract (except appendectomy)
7. History of relevant orthostatic hypotension, fainting spells or blackouts
8. Known hypersensitivity to any component of the formulation (telmisartan and hydrochlorothiazide), or to any other angiotensin II receptor blocker (ARBs), any other thiazides, or thiazide derivatives (e.c. sulfonamide derivatives like a chlorthalidone)
9. Intake of drugs with a long half-life (≥24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 7 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within 4 months or 6 half-lives of the investigational drug prior to administration
12. Smoker (≥20 cigarettes/day)
13. Alcohol abuse (60 g or more ethanol/day: ex. 3 middle-sized bottles of beer, 3 gous (equivalent to 540 mL) of sake)
14. Drug abuse
15. Blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
16. Excessive physical activities (within 1 week prior to administration or during the trial)
17. Intake of alcohol within 2 days prior to administration
18. Inability to comply with dietary regimen of study centre
19. Inability to refrain from smoking on trial days
20. Subjects judged to be inappropriate by the investigator or the sub-investigator

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in the plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) | Up to 72 hours after drug administration
The maximum measured concentration of the analyte in the plasma (Cmax) | Up to 72 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in the plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 72 hours after drug administration
Time from dosing to the maximum concentration of the analyte in the plasma (tmax) | Up to 72 hours after drug administration
Terminal rate constant in the plasma (λz) | Up to 72 hours after drug administration
Terminal half-life of the analyte in the plasma (t1/2) | Up to 72 hours after drug administration
Mean residence time of the analyte in the body after oral administration (MRTpo) | Up to 72 hours after drug administration
Number of participants with abnormal findings in physical examination | Up to 72 hours after drug administration
Number of participants with clinically significant findings in vital signs | Up to 72 hours after last drug administration
Number of participants with clinically significant findings in 12-lead ECG | Up to 72 hours after drug administration
Number of participants with clinically significant findings in clinical laboratory parameters | Up to 72 hours after drug administration
Number of participants with adverse events | Up to 7 days after drug administration